CLINICAL TRIAL: NCT05751603
Title: Comparison of Smooth Emergence During Extubation After Anesthesia When Sugammadex is Administered Before and After Extubation
Brief Title: Effectiveness on Smooth Extubation According to the Administration Time of Sugammadex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJOUIRB-INT-2022-173
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Sugammadex; Extubation; Smooth Emergence
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Routine anesthetic process; sugammadex is administered when spontaneous respiration is returned (before extubation)
- Experimental group (Experimental): sugammadex is administered just after extubation.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — sugammadex is administered just after extubation
  Arms: Experimental group

SUMMARY:
After surgery is completed under general anesthesia, extubation is performed after recovery from anesthesia, and during this process, bucking, coughing, and rapid and excessive hemodynamic fluctuations occur very often. These phenomena can lead to high intrathoracic pressure, venous congestion, hematoma formation, or increased bleeding after major neck surgery. (1) They can also increase the risk of aerosol generation, which can transmit infection to health care workers. (2) For this, smooth extubation is required. Methods of administering drugs such as lidocaine, opioids, or dexmedetomidine have been proposed for smooth extubation. (3-5) As a disadvantage, the use of these drugs may be associated with deep sedation and reduced airway reflexes .

Recently, Babu et al. (6) reported that bucking and coughing during extubation could be reduced by changing the timing of administering a muscle relaxant antagonist rather than using these sedative drugs, and thus complications related to extubation could be reduced. In general, in the awakening process, it was common to administer the muscle relaxant at the point of recovery of spontaneous breathing. However, Babu et al. demonstrated the possibility of safe and smooth extubation by changing the timing of administering neostigmine without the use of sedatives or narcotic analgesics, but there are few studies on sugammadex.

Therefore, when recovering from general anesthesia, sugammadex was administered before and immediately after extubation to evaluate and compare smooth extubation (ie, comparison of the frequency of bucking and coughing).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia for thyroid surgery.
* aged between 19 and 64 years
* American Society of Anesthesiologists physical status I and II

Exclusion Criteria:

* patients with malformation or tumor of the upper respiratory tract
* patients with risk of aspiration
* obese cases with a BMI > 35
* patients in which tracheal intubation was difficult
* refusal to participate in research

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-03 (Estimated); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
extubation quality score | immediate after extubation
  score based on the incidence and severity of coughing straining

SECONDARY OUTCOMES:
time to respiration | immediate after extubation
  time from withdrawal of anesthetics to respiration
time to extubation | immediate after extubation
  time from withdrawal of anesthetics to extubation
sore throat in postanesthetic care unit | in postanesthetic care unit
  Scores obtained by questioning the patient in postanesthetic care unit

IPD SHARING:
Plan to Share IPD: Undecided